CLINICAL TRIAL: NCT04482049
Title: A Prospective, Multicenter, Non-interventional Study to Investigate the Disease Characteristics of Adult Patients With Long Chain Fatty Acid Oxidation Disorders (FAOD)
Brief Title: A Prospective Study of the Disease Characteristics of Adult Patients With Long Chain Fatty Acid Oxidation Disorders
Acronym: FORWARD
Status: Completed | Type: Observational
Sponsor: Reneo Pharma Ltd (Industry)
Responsible Party: Sponsor
Organization: OnKure, Inc. (Industry)
Other Study IDs: REN001-903
Record Dates: First submitted 2020-07-14; First posted 2020-07-22 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Fatty Acid Oxidation Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to collect information on disease characteristics from adult patients diagnosed with fatty acid oxidation disorders (FAOD).

DETAILED DESCRIPTION:
In this study there will be no drug intervention. The study will include a Baseline visit and a follow up visit scheduled at Month 4. At these visits medical history, safety assessments, concomitant medications, exercise tests and quality of life questionnaire data will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. A genetically confirmed diagnosis of one of the following:

   1. Carnitine palmitoyltransferase 2 deficiency
   2. Very long-chain Acyl-CoA dehydrogenase deficiency
   3. Long-chain 3-hydroxyacyl-CoA dehydrogenase deficiency
   4. Trifunctional protein deficiency
2. A stable treatment regimen for at least 30 days
3. Ambulatory and able to perform the study exercise test, using walking aids if necessary
4. Willing and able to personally sign and date an informed consent document indicating that the subject has been informed of all pertinent aspects of the study

Exclusion Criteria:

1. Unstable or poorly controlled disease as determined by one or more of the following:

   1. Presence of symptoms of acute rhabdomyolysis with clinically significant elevations in serum CK
   2. Evidence of acute crisis from their underlying disease
2. Currently taking a PPAR agonist
3. Have motor abnormalities other than those related to the fatty acid oxidation disorder that could interfere with the study procedures, as determine by the investigator
4. Evidence of significant concomitant medical or psychiatric disease that in the opinion of the Investigator may interfere with the conduct or safety of this study
5. Pregnant or nursing females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from centres experienced in the identification and subsequent management of patients with long chain FAOD.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
To evaluate change in function as measured by 12 minute walk test in adult subjects with long chain FAOD | Week 16
  Change from baseline in 12MWT

SECONDARY OUTCOMES:
To evaluate change in symptoms related to FAOD using a newly developed muscle symptom questionnaire specifically designed for adult patients with long chain FAOD | Week 16
  Change from baseline in FAOD-Muscle Symptom Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Gillingham, PhD, RD, LD, Principal Investigator — Dept of Molecular and Medical Genetics, Oregon Health and Science University
Locations (15):
- United States (3):
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbuilt University Medical Center, Nashville, Tennessee
- Medizinische Universität Innsbruck, Innsbruck, Austria
- UZ Leuven University Hospitals Leuven, Leuven, Belgium
- Vseobecna fakultni nemocnice v Praze, Klinika pediatrie a dedicnych poruch metabolizmu, Prague, Czechia
- Rigshospitalet, Klinik for nerve- og muskelsygdomme, Copenhagen, Denmark
- Hôpital Pitié-Salpêtrière, Paris, France
- Pest Megyei Flór Ferenc Kórház, Kistarcsa, Hungary
- Italy (2):
  - Universita di Brescia, Brescia
  - Azienda Ospedaliera Universitaria Policlinico "G. Martino" di Messina, Messina
- Uniwersyteckie Centrum Kliniczne, Gdansk, Poland
- Spain (2):
  - Hospital 12 de Octubre, Madrid
  - Unidad de Diagnóstico y Tratamiento de Enfermedades Metabólicas Complejo Hospitalario Universitario de Santiago Travesía de Choupana s/n, Santiago de Compostela
- Salford Royal NHS Trust, Salford, United Kingdom